CLINICAL TRIAL: NCT05973422
Title: Sigi Insulin Management System - First-in-Human Study
Brief Title: Sigi Insulin Management System - A First-in-Human Study in Adults With Type 1 Diabetes
Acronym: SigiFIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-0001 Sigi FIH Study CIP
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
Keywords: Insulin patch pump; CGM control; Smartphone control; Pre-filled insulin cartridges; Occlusion detection
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIGI Insulin Management System Observed and At-Home Use (Experimental): Current insulin pump users with type 1 diabetes, age 18+, will use the SIGI insulin management system for 1 day observed in the hospital setting, then for 2 more weeks of outpatient use.
  Interventions: Device: SIGI Insulin Management System

INTERVENTIONS:
Device: SIGI Insulin Management System — Continuous subcutaneous insulin infusion with Sigi, and wearing the Dexcom G7 sensor using the Dexcom App.

SUMMARY:
This early feasibility first-in-human study is a prospective single-arm single-center study of Sigi insulin patch pump. After a 1st day and night under medical surveillance during a hotel stay, Sigi system will be evaluated during 15 days at home in adults with type 1 diabetes.

DETAILED DESCRIPTION:
Sigi Insulin Management System (Sigi) is a novel insulin patch pump intended for subcutaneous delivery if insulin at set and variable rates for the management of diabetes mellitus in persons requiring insulin. Sigi is offering superior delivery accuracy and precision, accelerated occlusion detection, wearable patch pump, pre-filled insulin cartridges and smartphone control.

Glycemia is CGM controlled and for safety purposes, CGM data are shared with study medical team during the whole study.

Sigi FIH Study is conducted in a single clinical site in Lausanne University Hospital (CHUV) in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients with T1D since more than 1 year
* Adults 18+years
* Patients under sensor augmented pump for at least 6 months
* Hybrid closed-loop users willing to switch to manual mode 15 days before study
* Patients with calculated insulin-to-carb ratio and correction factor
* Patients with total daily insulin above 30 insulin units
* Patients with correction factor below 3.5 mmol/L
* No severe hypoglycemic or ketoacidosis episode requiring third-party intervention within the past 12 months
* Active users of Teflon infusion sets
* Patients willing to use a smartphone interface to use their pump and to answer study questionnaires

Exclusion Criteria:

* Patients with T2D
* Patients with T1D under multiple daily injections
* Patients using Apidra and not willing to switch to NovoRapid / Fiasp / Humalog
* Patients with history of skin diseases (e.g. generalized eczema, plan lichen, psoriasis)
* Patients with known allergy to some insulins
* Clarke's score ≥ 4 (hypoglycemia unawareness)
* Severe late complications of diabetes, like severe neuropathy, non-stabilized proliferative retinopathy, EGF < 30 mL/min, myocardial infarction or stroke within the last 3 months
* Glycated hemoglobin HbA1c > 8.5 % at screening visit
* Medications interacting with glucose homeostasis (e.g. steroids)
* Pregnant of breastfeeding women
* Planned operation / MRI / CT requiring removal of infusion pad over the 15 days of the study
* Planned travel over the 15 days of the study
* Persons under guardianship or incapable of judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 15 days
  Number of serious adverse events
Adverse Events | 15 days
  Number of adverse events
Adverse Device Effects | 15 days
  Number of adverse device effects (ADE)
Serious adverse device effects (SADE) | 15 days
  Number of serious adverse device effects (ADE)

SECONDARY OUTCOMES:
Severe hypoglycemia events, as a indicator of successful CSII self-management with Sigi | 15 days
  Number of severe hypoglycemia events (with cognitive impairment such that assistance of another individual is needed for treatment) during study
Diabetic ketoacidosis events, as a indicator of successful CSII self-management with Sigi | 15 days
  Number of diabetic ketoacidosis events
Acceptance and confidence of PI to proceed to outpatient use | 1 day
  Number of participants who pass the observed use setting as evaluated by PI and proceed to outpatient use.
Acceptance and confidence of participant to proceed to outpatient use | 1 day
  Number of participants who pass the observed use setting as evaluated by participants and proceed to outpatient use.
Device deficiencies | 15 days
  Number of device deficiencies (device issues) recorded during study use
Evaluation of pad duration (days) | 15 days
  Collect pad replacement dates to calculate the pad survival rate at 3 days
Occlusion detection rate | 15 days
  Rate of occlusions detected by the system over the total wear period (number of occlusions/total wear time in days)
Evaluation of skin tolerance | 15 days
  Number of recorded skin reactions, including skin related adverse events, during the 15 day wear time.
Evaluation of overall device tolerance | 15 days
  Number of reports related to discomfort at the infusion site, including discomfort related adverse events, during the 15 day wear time.
System Usability Scale (SUS) at baseline and 15 days for the PAD | 15 days
  System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicating better perceived usability, collected at baseline and 15 days for evaluation of the PAD.
System Usability Scale (SUS) at baseline and 15 days for the Pump Assembly | 15 days
  System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicating better perceived usability, collected at baseline and 15 days for evaluation of the pump assembly.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Wojtusciszyn, MD, Principal Investigator — CHUV Centre Hospitalier Universitaire Vaudois

IPD SHARING:
Plan to Share IPD: No